CLINICAL TRIAL: NCT05464927
Title: Visualizing Vascular Mechanisms of Lipedema
Acronym: VMP
Status: Active, not recruiting | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Rachelle Crescenzi, Associate Professor, University of Virginia
Other Study IDs: 302197; 1R01HL157378-01 (NIH); 210181 (Other: Vanderbilt University Medical Center)
Record Dates: First submitted 2022-07-08; First posted 2022-07-19 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Lipedema
Keywords: MRI; Sodium; Adipose Tissue; fibrosis; lipedema
MeSH Terms: conditions — Lipedema; Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples obtained during the course of this research will be aliquoted, de-identified and stored in freezers for future analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Participants pre CDT: * Participants with lipedema
  * Biologically Female
  * Age range = 18-80 years
  * BMI range = 18 to 40 kg/m2
  * BMI range = 18 to 40 kg/m2
- Controls: * Participants without lipedema
  * Biologically Female
  * Age range = 18-80 years
  * BMI range = 18 to 40 kg/m2
- Participants post CDT: * Participants with lipedema
  * Biologically Female
  * Age range = 18-80 years
  * BMI range = 18 to 40 kg/m2
  * BMI range = 18 to 40 kg/m2

SUMMARY:
This work will address clinical unmet needs for patients with lipedema using advanced magnetic resonance imaging (MRI) methods, in sequence with portable clinical tools, by testing fundamental hypotheses regarding potential screening methods, lymphatic therapy, and vascular dysfunction in patients with lipedema.

DETAILED DESCRIPTION:
Lipedema is a disease marked by disproportionate subcutaneous adipose tissue (SAT) accumulation in the lower extremities that is accompanied by somatic pain and edema. Importantly, lipedema is commonly misdiagnosed as obesity and has been estimated to affect a high 11% of women. However, symptoms are refractory to diet, exercise, and other interventions for obesity leading to a mean delayed diagnosis of 22 years, high physical morbidity, and lifelong distress. Despite growing awareness of lipedema as a distinct clinical entity and a recent call to action for lipedema research, fundamental gaps persist in knowledge regarding both disease mechanisms and treatment options for this debilitating disease.

Over the past four years, multi-disciplinary study from investigators in radiology, vascular medicine, and physical therapy has demonstrated that lipedema has distinct characteristics from obesity. Using whole-body fat-and-water MRI, lipedema is characterized by a 42% higher lower-extremity SAT deposition compared to BMI-matched females without lipedema (p<0.001). Using noninvasive sodium MRI technologies, skin sodium is also elevated in patients with lipedema compared to controls (14.9±2.9 vs. 11.9±2.0 mmol/L, p=0.01) in the lower extremities, but not upper extremities. Importantly, skin sodium decreases following 6-weeks of lymphatic stimulation by complete decongestive therapy (CDT) in preliminary study of patients with lipedema. These tissue signatures are consistent with those of patients with known lymphatic insufficiencies (i.e., secondary lymphedema). Recent findings of elevated arterial perfusion and inflammatory profiles in lipedema raise significant questions about how blood and lymphatic circulation are involved in lipedema.

The critical barrier to interrogating these systems, and more broadly addressing clinical unmet needs for evidence-based therapies for patients with lipedema, is that noninvasive lymphatic imaging strategies are traditionally underdeveloped. To address this barrier, non-tracer based MR lymphangiography is capable of visualizing lymphatic dilation and stasis in unilateral lymphedema, and similar features of lymphatic insufficiency are observed in the lower extremities of patients with lipedema.

This study will apply these MRI tools together with standard clinical tools to test the following hypotheses:

Hypothesis 1A: Ultrasound can be used as an accessible alternative to MRI for measuring subcutaneous fat deposition to distinguish lipedema from obesity.

Hypothesis 1B: Ultrasound measurement of fat deposition together with bedside tools for measuring water deposition have improved ability than ultrasound alone for distinguishing lipedema from controls.

Hypothesis 2: Tissue sodium is reduced following CDT in the lower extremities, but not in the untreated upper extremities, of patients with lipedema consistent with improved patient-reported outcomes.

Hypothesis 3: Lymphatic flow velocity is reduced, while arterial blood flow is elevated, in the legs of patients with lipedema compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* Participants with and without lipedema
* Biologically Female
* Age range = 18-80 years
* BMI range = 18 to 40 kg/m2

Exclusion Criteria:

* Primary lymphedema
* Contraindication to 3T MRI
* Pregnant
* Severe claustrophobia
* Inability to provide written, informed consent
* Active infection anywhere in the body, or open wound on the lower-extremities or at locations for measurement

Also excluded are subjects incapable of giving informed written consent:

* Subjects who have an inability to communicate with the researcher for any reason
* Subjects who are non-English speaking who cannot communicate through a translator, or if a translator is not available
* Subjects who cannot adhere to the experimental protocols for any reason
* Subjects who have limited mental ability to give informed consent due to mental disability, confusion, or psychiatric disorders
* Prisoners

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study Population:
  The investigators will recruit adults with and without lipedema
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in tissue sodium content: quantification of tissue sodium content in treated limbs following the completion of therapy | at baseline and approximately 6 weeks later
  Tissue sodium content (mmol/L) quantified by sodium MRI
Change in lymphedema severity: quantification of lymphatic stasis in treated limbs following the completion of therapy | at baseline and approximately 6 weeks later
  Lymphatic stasis area (mm^2) quantified by MR lymphangiography
Baseline tissue sodium content: quantification of tissue sodium in affected limbs | At baseline
  Tissue sodium content (mmol/L) quantified by sodium MRI
Baseline lymphedema severity: quantification of lymphatic stasis in affected limbs | At baseline
  Lymphatic stasis area (mm^2) quantified by MR lymphangiography
Change in limb extracellular water: quantification of limb extracellular water in treated limbs following the completion of therapy | at baseline and approximately 6 weeks later
  Limb extracellular water (Ohms) estimated by bioimpedance spectroscopy
Change in skin water: quantification of skin water in treated limbs following the completion of therapy | at baseline and approximately 6 weeks later
  Skin water (percent) estimated by tissue dielectric probe
Change in skin elasticity: quantification of skin elasticity in treated limbs following the completion of therapy | at baseline and approximately 6 weeks later
  Skin elasticity (Newtons) quantified by fibrometer
Baseline limb extracellular water: quantification of limb extracellular water in affected limbs | At baseline
  Limb extracellular water (Ohms) estimated by bioimpedance spectroscopy
Baseline skin water: quantification of skin water in affected limbs | At baseline
  Skin water (percent) estimated by tissue dielectric probe
Baseline skin elasticity: quantification of skin elasticity in affected limbs | At baseline
  Skin elasticity (Newtons) quantified by fibrometer

CONTACTS AND LOCATIONS:
Overall Officials: Rachelle Crescenzi, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided